CLINICAL TRIAL: NCT00635401
Title: A Multicenter, Open-Label Study Exploring the Efficacy and Safety of Varenicline in Japanese Smokers Motivated to Quit Smoking
Brief Title: A Study of the Efficacy and Safety of Varenicline in Japanese Smokers Motivated to Quit Smoking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3051043
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.5 mg BID (Experimental)
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — 0.5 mg BID for 7 weeks
  Other Names: Chantix, Champix, CP-526,555

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of varenicline in Japanese smokers. Efficacy is evaluated by continuous quit rate and withdrawal symptoms of smokers. Safety is evaluated by adverse events, laboratory tests, and other safety tests.

ELIGIBILITY:
Inclusion Criteria:

* Japanese smokers motivated to quit smoking
* No period without smoking of more than 3 months
* Smoked an average of at least 10 cigarettes/day in the past year

Exclusion Criteria:

* Subjects who have used nicotine replacement therapy within 1 month of the study screening visit
* Subjects intending to use nicotine replacement therapy or other smoking cessation treatments during the study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-05; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Carbon monoxide (CO)-confirmed 4-week continuous quit rate (4-week CQR) from Weeks 4 to 7. | Weeks 4-7

SECONDARY OUTCOMES:
CO-confirmed 7-day Point Prevalence from Week 2 through Week 7. | Weeks 2-7
Continuous abstinence rate from target quit date (TQD) from Week 2 through Week 7. | Weeks 2-7
Average number of daily cigarettes smoked from Week 2 through Week 7. | Weeks 2-7
Assessment of withdrawal symptoms by Minnesota Nicotine Withdrawal Scales (MNWS) from Week 2 through Week 7. | Weeks 2-7
Assessment of satisfaction (desirable and aversive effects) obtained from smoking by Smoking Effects Inventory (SEI) (administered only to subjects who had smoked since the previous assessment) from Week 2 through Week 7. | Weeks 2-7
Assessment of tobacco craving by the Brief Questionnaire of Smoking Urges (QSU-Brief) from Week 2 through Week 7. | Weeks 2-7
Assessment of the effect of smoking cessation on subjects' quality of life by the Smoking Cessation Quality of Life (SCQoL) questionnaire from Week 2 through Week 7. | Weeks 2-7
Adverse events, laboratory test changes throughout the study. | Weeks 1-7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Japan (8):
  - Pfizer Investigational Site, Chuo-ku Fukuoka, Fukuoka
  - Pfizer Investigational Site, Nishi-ku Yokohama, Kanagawa
  - Pfizer Investigational Site, Beppu, Oita Prefecture
  - Pfizer Investigational Site, Ōita, Oita Prefecture
  - Pfizer Investigational Site, Hamamatsu, Shizuoka
  - Pfizer Investigational Site, Edogawa-ku, Tokyo
  - Pfizer Investigational Site, Minato-ku, Tokyo
  - Pfizer Investigational Site, Toshima-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051043&StudyName=A%20study%20of%20the%20efficacy%20and%20safety%20of%20varenicline%20in%20Japanese%20smokers%20motivated%20to%20quit%20smoking